CLINICAL TRIAL: NCT04613219
Title: Correlation Between the Change of Peripheral Lymphocyte Subsets and Clinically Amyopathic Dermatomyositis Combined With Rapidly Progressive Interstitial Lung Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jing Liang (Other)
Responsible Party: Sponsor-Investigator, Jing Liang, dean of orthopedic department, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: TY017AN
Record Dates: First submitted 2020-09-15; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-09

CONDITIONS: Clinically Amyopathic Dermatomyisitis(CAMD)
MeSH Terms: interventions — tofacitinib

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Tofacitinib 5 MG [Xeljanz] — Treatment with Tofacitinib

SUMMARY:
Acute respiratory distress syndrome (ARDS) occurs in Clinically Amyopathic Dermatomyisitis(CADM) combined with Rapidly Progressive Interstitial Lung Disease(RPILD) within 1-3 months, which leads to death of patients and is difficult to treat. Even if high doses of glucocorticoids are ineffective, there is no recommended treatment for such patients, which is a huge medical challenge.Lymphopenia is an independent risk factor for death in CADM-RPILD, but the cause of lymphopenia is unclear.In this study, the level of lymphocyte subsets in peripheral blood was detected by flow cytometer, in order to further clarify the pathogenesis of the disease, to facilitate clinical guidance of treatment, and to improve the survival rate of patients.In addition, studies have shown that INF-α levels are significantly increased in CADM patients combined with RPILD and are a poor prognostic factor for CADM-RPILD, suggesting that the interferon system plays a role in the pathogenesis of CADM and can be used as an evaluation index of the severity of CADM-RPILD.In this study, the levels of relevant cytokines including INF and IL-2, IL-17, IL-18, IL-6 were detected simultaneously, and the relationship between disease activity and lymphocyte subsets was analyzed, and the changes of lymphocyte subsets after Tofacitinib treatment were determined in order to facilitate clinical guidance of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years old,≤80years old,no gender limit;
2. CADM of diagnosis according to Sontheimer diagnostic criteria;
3. combined with Rapidly Progressive Interstitial Lung Disease

Exclusion Criteria:

1. Age<18years old，>80years old;
2. potential malignant tumor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with Clinically Amyopathic Dermatomyisitis combined with Rapidly Progressive Interstitial Lung Disease
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
The level of a lymphocyte in a lymphocyte subset correlates with disease activity. | 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- Qianfoshan Hospital, Jinan, Shandong, China